CLINICAL TRIAL: NCT05457166
Title: Interest in Using the KASPARD System for the Prevention of Falls in Nursing Homes (EHPAD, for Its French Acronym)
Brief Title: Use of the KASPARD System for Fall Prevention in Nursing Homes
Acronym: KASPARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020_89; 2021-A03210-41 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-06

CONDITIONS: Accidental Falls; Nursing Homes
Keywords: Elderly person; EHPAD; Fall; Prevention; Detection system
MeSH Terms: interventions — Home Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental): patients in a before/after experimental design to assess the value of using the KASPARD technology compared to the conventional management of patients with falls in nursing homes
  Interventions: Device: KASPARD system for fall prevention in nursing homes

INTERVENTIONS:
Device: KASPARD system for fall prevention in nursing homes — All subjects will be monitored for 2 periods of 100 nights each. Recordings will be made continuously at night for the duration of the study Period 0: set-up, adjustment, recording (without alarm); This is a preparatory phase which is part of the usual use of the device.
  Duration: 10 days Before period: The BEFORE period runs for 100 nights during which the device alarm is not activated, but the device records events.
  After period: The AFTER period is 100 nights during which the device alarm is activated: Monitoring with recording + alarm activated (usual care + action if alarm is triggered)

SUMMARY:
Falls are a frequent cause of admission to nursing homes [2]. It is also the most frequently reported adverse event in these institutions.

The prevention of falls in EHPAD must mobilise several levers of action and involve all staff. It must be included in the establishment's project in the same way as the policy on the proper use of restraints [21].

Home automation and new technologies can contribute to the prevention of falls and their consequences. Most of the existing solutions on the market are either fall detection solutions based on a watch or pendant or rise detection solutions based on a sub-mattress or floor mat. All of these solutions work with a contact and often require a daily set-up or check by the care teams. But the real challenge today for new technologies is to prevent falls in the elderly, by directly addressing the risk factors.

KASPARD is a non-contact (remote sensors) and non-intrusive (no video image, it uses point cloud technology) solution for detecting falls, excessive wandering and nocturnal activities in a nursing home. The information is transmitted securely via the wifi network to a mobile phone (or TSI/DECT) and to a computer. The KASPARD solution, which is already on the market (non-medical CE marking), is used in several EHPADs in Belgium and France. It is not a medical device. To date, it has a sensitivity and specificity of over 90% (manufacturer's unpublished data).

We wish to verify the effectiveness of the KASPARD technology for the prevention of falls in EHPAD, suggested for the moment by an observational study, with the help of a multi-centre clinical study

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female resident of an EHPAD
* Person aged ≥ 65 years
* Elderly person at high risk of falling (fell at least 1 time in the 6 months prior to inclusion)
* Resident or his/her legal representative who has given free, written, informed consent to participate in the trial
* Socially insured resident
* Resident willing to comply with all study procedures and duration. The questionnaires used will be validated questionnaires for the target population (QoL-AD questionnaire for residents and their carers).

Exclusion Criteria:

* Refusal to participate in the study
* Elderly resident who has a fall and for whom the use of a restraint is deemed essential by the coordinating doctor of the EHPAD
* Persons under legal protection are not excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
the number of falls observed over a period of 100 nights with KASPARD | 100 nights
  To show that the KASPARD system reduces the number of falls observed over a period of 100 nights with the device activated compared to a period of 100 nights with the device deactivated, in elderly people aged over 65 years residing in EPAD and at high risk of falling.

SECONDARY OUTCOMES:
The number of night shift interventions | 100 nights with the device on versus 100 nights with the device off
The number of nights without restraint | 100 nights with the device on versus 100 nights with the device off
The time taken to intervene after a fall | 100 nights with the device on versus 100 nights with the device off
  Time between the occurrence of the fall and the arrival of staff at the patient's bedside
Fear of falling assessed by the FES scale | 100 nights with the device on versus 100 nights with the device off
  Fear of falling reported by residents at the end of each period: last day of period 1 and last day of period 2
Quality of life questionnaire | 100 nights with the device on versus 100 nights with the device off
  Quality of life questionnaire reported by the patient and once at the end of each period: last day of period 1 and last day of period 2
Resident satisfaction | activation period of 100 nights
  Resident satisfaction will be assessed by a satisfaction questionnaire
Night and day staff satisfaction | activation period of 100 nights
  Staff satisfaction will be assessed by a satisfaction questionnaire evaluating organisational aspects, disturbance of walking patients, interest in the reports provided by the system

CONTACTS AND LOCATIONS:
Overall Officials: François Puisieux, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Pôle de gérontologie - Hôpital Les Bateliers, Lille, France